CLINICAL TRIAL: NCT06604819
Title: The Impact of Ozone Gel on the Bone Height and Density After Closed Sinus Lifting with Simultaneous Implant Placement: a Randomized Controlled Clinical Trial.
Brief Title: The Impact of Ozone Gel on the Bone Height and Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Dina yousry, Principle investigator "Doctorate candidate", Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 417/2021
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Sinus Pneumatization
Keywords: closed sinus lifting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: biostatistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- closed sinus lifting using osteotomes with simultaneous implant placement (Active Comparator): Full thickness mucoperiosteal flap was elevated.• The pilot drill of the implant system was used to create an osteotomy 1 mm short of the subantral floor. • The insertion of the osteotome were repeated several times until the required membrane lift was achieved then the osteotome corresponding in size to the last drill was used.After that, placement of the implant was done .Healing abutment was placed to allow for multiple times measurements of implant stability and primary closure was done and the flap was sutured in an interrupted manner using 4/0 prolene suture .
  Interventions: Procedure: closed sinus lifting using osteotomes with simultaneous implant placement
- closed sinus lifting using osteotomes with simultaneous implant placement with ozone gel placement (Experimental): Full thickness mucoperiosteal flap was elevated.• The pilot drill of the implant system was used to create an osteotomy 1 mm short of the subantral floor. • The insertion of the osteotome were repeated several times until the required membrane lift was achieved then the osteotome corresponding in size to the last drill was used.Ozone gel was delivered into the osteotomy . To obtain the ozone gel, pure olive oil was blasted with 25 μ/ml O3 gas for two days, or until the oil changed from a greenish-colored liquid to a whitish gel. The longevity Ext 120 ozone generator executed out this process. After that, placement of the implant was done .Healing abutment was placed to allow for multiple times measurements of implant stability and primary closure was done and the flap was sutured in an interrupted manner using 4/0 prolene suture .
  Interventions: Drug: Ozone gel placed after closed sinus lifting then implant placed simultaneously.

INTERVENTIONS:
Drug: Ozone gel placed after closed sinus lifting then implant placed simultaneously. — The patient received closed sinus lifting using osteotomes then ozone gel is prepared. Pure olive oil was blasted with 25 μ/ml O3 gas for two days, or until the oil changed from a greenish-colored liquid to a whitish gel. The longevity Ext 120 ozone generator executed out this process then implants were placed.
  Arms: closed sinus lifting using osteotomes with simultaneous implant placement with ozone gel placement
Procedure: closed sinus lifting using osteotomes with simultaneous implant placement — The patient received closed sinus lifting using osteotomes with implant placed simultaneously.
  Arms: closed sinus lifting using osteotomes with simultaneous implant placement

SUMMARY:
Purpose: The present study was conducted to evaluate the effect of using ozone gel with maxillary sinus elevation using tenting technique on the clinical and radiographic outcome of implants placed simultaneously..

Materials and Methods: A total of 30 sinuses with an average residual alveolar bone height ranging from 4-7 mm participated in this randomized controlled clinical trial. After closed sinus lift operation, patients were randomly and equally allocated into control group and ozone gel recipient group. Cone beam computed tomography was performed immediately and at 4 months postoperatively. Bone stability was measured immediately and at 3 & 4 months postoperatively. Bone height and stability were evaluated radiographically, and bone stability was measured using the Osstell device.

DETAILED DESCRIPTION:
Concern over biological augmentations used in bone healing has grown in recent years. One of the essential demands in sinus lifting procedure is to speed up the bone formation and enhance the quality of the formed bone in the space created after sinus elevation. Since more than 100 years medical grade ozone has been used as one of the non-medication methods of treatment. E. A. Fisch in the 1930's was the first dentist to use ozone therapy in his practice to aid in disinfection and wound healing. Current ozone uses a mixture of ozone gel and pure oxygen, with today's medical ozone generators which regulate the flow of medical grade O2 through high voltage tubes which is capable of producing pure ozone-oxygen mixtures in precise dosages.

Nevertheless, there is not enough evidence to support the use of ozone in oral and maxillofacial surgery. Ozone therapy has a therapeutic effect that promotes blood and growth factor supply, aids in wound healing, and may improve bone regeneration . However up till now, no studies were conducted to assess the impact of using ozone gel on bone formation in case maxillary sinus elevation.

ELIGIBILITY:
Inclusion Criteria:

* Patient age should be > 18 years of age.
* Patients included were ASA I and ASA II.
* Both males and females were included in the study.
* Patients with need of tooth replacements in the maxillary premolar and molar area where the residual alveolar bone height ranges from 4-7 mm and bone density D3 or D4.
* Compliance with all requirements in the study and signing the informed consent.

Exclusion Criteria:

* Patients with immunological diseases or diseases affecting bone healing.
* Patients suffering from uncontrolled systemic diseases.
* Patients with active acute infection related to the planned implant site, maxillary sinusitis or pathosis.
* Patients with parafunctional occlusal habits.
* Patients with bad oral hygiene.
* Patients who were alcohol and drug abusers.
* Heavy Smoker Patients.
* Patients who went previous sinus lifting surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Implant stability | Immediate postoperative,3 months and 4 months postoperative
  - Resonance frequency analysis was performed to assess implant stability. The implant stability was measured using the Osstell ISQ scale "immediate postoperative then after 3 and 4 months . The readings were taken along the three surfaces of the implant (perpendicular to the implant axis, mesial surface and distal surface). Finally, the averages of these readings were taken as a representative value for each implant .

SECONDARY OUTCOMES:
Bone Density | Immediate postoperative and 4 months postoperative
  The bone density was evaluated using CBCT. To minimize the error from radiographic image alignment, the On Demand 3D fusion module software was used to generate a superimposed image at the sagittal and coronal planes of each implant to compare each parameter .
Bone height gain | Immediate postoperative and 4 months postoperative
  Cone beam computed tomography (CBCT was taken to evaluate the accuracy of implant placement and to represent the baseline measurement for evaluation. The bone height gain was evaluated along the surface of each implant.

CONTACTS AND LOCATIONS:
Overall Officials: Dina El-Zaefzaf, Masters, Principal Investigator — Suez Canal University
Locations (1):
- Faculty of Dentistry, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
It will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It will be available after the research is published.
Access Criteria: It will be available upon request

REFERENCES:
- [Derived] Yousry D, Riad R, Soliman RA, ElSholkamy M. Does ozone gel enhance the bone width and buccal plate of bone thickness surrounding the implant following osseodensification? A randomized controlled clinical trial. Oral Maxillofac Surg. 2025 Apr 14;29(1):82. doi: 10.1007/s10006-025-01367-x. PMID 40229413